CLINICAL TRIAL: NCT01005264
Title: Effectiveness of Removable Walker Cast Versus Non-removable Fiberglass Off-bearing Cast in the Healing of Diabetic Plantar Foot Ulcer- a Randomized Controlled Trial
Brief Title: Removable Walker for Neuropathic Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Multimedica (Other)
Responsible Party: Ezio Faglia MD, Diabetic Foot Center - IRCCS Multimedica, Sesto San Giovanni (Milan), Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2007cardiovascolare
Record Dates: First submitted 2009-10-19; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; neuropathic plantar ulcer; ulcer healing; non-removable total contact cast; removable cast walker
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-removable fiberglass (Active Comparator): Softcast3M®, 3M Health Care, St. Paul, MN (USA) were used for construction of the pressure-relief apparatus
  Interventions: Device: non-removable fiberglass
- Stabil-D® (Active Comparator): Composed of a specifically designed rigid, boat shaped, and fully rocker bottom sole
  Interventions: Device: Stabil-D®

INTERVENTIONS:
Device: non-removable fiberglass — Two types of fiberglass bandages (Softcast3M®, 3M Health Care, St. Paul, MN (USA)) were used for construction of the pressure-relief apparatus
  Other Names: Softcast3M®, 3M Health Care, St. Paul, MN (USA)
  Arms: non-removable fiberglass
Device: Stabil-D® — Stabil-D Stabil-D® is composed of a specifically designed rigid, boat shaped, and rocker sole
  Other Names: Podartis srl, Montebelluna, Treviso, Italy
  Arms: Stabil-D®

SUMMARY:
1. Objective: To evaluate the efficacy of removable cast walker compared to non-removable fiberglass off-bearing cast in the treatment of diabetic plantar foot ulcer
2. Research design and methods: Forty-five adult diabetic patients with non-ischemic, non-infected neuropathic plantar ulcer were randomized to treatment with a non-removable fiberglass off-bearing cast (TCC group) or walker cast (Stabil-D group). Treatment duration was 90 days. Percent reduction in ulcer surface area and total healing rates were evaluated after treatment.

DETAILED DESCRIPTION:
Study design:

Two centers specializing in diabetic foot management (located in Sesto S. Giovanni and Milan, Italy) participated to this open, randomized clinical trial. The ethics-committee approved the study on January 10th, 2008. Enrollment of consecutive patients began February 2008 and ended March 2009. Eligible patients were fully informed of the study aim and procedures and written consent was obtained prior to study participation. Patients were then randomly assigned to one of the two treatment groups by opening randomization codebreak envelopes containing one of the two options. Separate randomization was performed for each center, and a copy of all randomization envelopes was kept at the statistical department of the Multimedica center. The two arms were composed of patients managed with non-removable fiberglass off-bearing cast (TCC group) and patients offloaded with the Stabil-D® (Podartis srl, Montebelluna, Treviso, Italy) walker cast (Stabil-D group).

ELIGIBILITY:
Inclusion Criteria:

* The presence of neuropathic plantar ulcer with an area graded IA according to the Texas University classification, AND
* The presence of peripheral neuropathy. Peripheral neuropathy was diagnosed based on insensitivity to a 10-g Semmes-Weinstein monofilament in more than 6 out of 9 areas of the foot and by a vibration perception threshold measured by biothesiometer (Neurothesiometer SLS, Nottingham, UK) at the malleolus > 25 volts.

Exclusion Criteria:

* Presence of an ankle-brachial pressure index (ABI) < 0.9 and/or transcutaneous oxygen tension (TcPO2) < 50 mmHg tested on the dorsum of the foot,
* Presence of clinical signs of infection, including edema, erythema, increased local skin temperature, or drainage,
* The probe-to-bone maneuver was required to be negative,
* Tthe standard X-ray examination of the foot was required to be negative for osteomyelitis,
* Use of steroids or cytostatic drugs,
* Presence of sensory, motor, or visual problems that could impair functional autonomy,
* Active ulcer on the contralateral foot,
* Previous major amputation of the contralateral limb,
* Previous or current deep venous leg thrombosis, OR
* Mental disorders interfering with patient compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Decrease in ulcer size | at 90th day

SECONDARY OUTCOMES:
Complete healing rate at the end of the study | at 90th day

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Faglia, MD, Principal Investigator — Diabetic Foot Center - IRCCS Multimedica, Sesto San Giovanni (Milan), Italy
Locations (1):
- Diabetic Foot Center - IRCCS Multimedica, Sesto San Giovanni, Milan, Italy

REFERENCES:
- [Result] Caravaggi C, Sganzaroli A, Fabbi M, Cavaiani P, Pogliaghi I, Ferraresi R, Capello F, Morabito A. Nonwindowed nonremovable fiberglass off-loading cast versus removable pneumatic cast (AircastXP Diabetic Walker) in the treatment of neuropathic noninfected plantar ulcers: a randomized prospective trial. Diabetes Care. 2007 Oct;30(10):2577-8. doi: 10.2337/dc07-0990. Epub 2007 Jun 11. No abstract available. PMID 17563333
- [Result] Piaggesi A, Macchiarini S, Rizzo L, Palumbo F, Tedeschi A, Nobili LA, Leporati E, Scire V, Teobaldi I, Del Prato S. An off-the-shelf instant contact casting device for the management of diabetic foot ulcers: a randomized prospective trial versus traditional fiberglass cast. Diabetes Care. 2007 Mar;30(3):586-90. doi: 10.2337/dc06-1750. PMID 17327325
- [Result] Caravaggi C, Faglia E, De Giglio R, Mantero M, Quarantiello A, Sommariva E, Gino M, Pritelli C, Morabito A. Effectiveness and safety of a nonremovable fiberglass off-bearing cast versus a therapeutic shoe in the treatment of neuropathic foot ulcers: a randomized study. Diabetes Care. 2000 Dec;23(12):1746-51. doi: 10.2337/diacare.23.12.1746. PMID 11128345
- [Derived] Faglia E, Caravaggi C, Clerici G, Sganzaroli A, Curci V, Vailati W, Simonetti D, Sommalvico F. Effectiveness of removable walker cast versus nonremovable fiberglass off-bearing cast in the healing of diabetic plantar foot ulcer: a randomized controlled trial. Diabetes Care. 2010 Jul;33(7):1419-23. doi: 10.2337/dc09-1708. Epub 2010 Mar 31. PMID 20357377